CLINICAL TRIAL: NCT01097577
Title: A Comparison of Pregabalin (Lyrica®) to Placebo in Postoperative Pain Relief of Patients Status-post Photorefractive Keratectomy: A Double-masked Randomized Prospective Study
Brief Title: A Comparison of Pregabalin (Lyrica®) to Placebo in Pain Relief After Photorefractive Keratectomy (PRK) Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Meek, Clinical Pharmacist, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20100004H
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
Keywords: photorefractive keratectomy; excimer laser; PRK; pain, postoperative; pregabalin
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregabalin (Experimental): Oral Pregabalin 75 mg capsule twice daily administered prior to PRK and continued for 5 days
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator): Oral placebo capsule (Lactose) twice daily administered prior to PRK and continued for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — 1 capsule (75 mg) by mouth twice daily starting two hours prior to surgery and continuing 4 days postoperatively.
  Other Names: Lyrica
  Arms: pregabalin
Drug: Placebo — 1 capsule by mouth twice daily starting two hours prior to surgery and continuing 4 days postoperatively.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of pregabalin to placebo for postoperative pain control after photorefractive keratectomy.

DETAILED DESCRIPTION:
Study subjects will be taken from a standard group of typical candidates for PRK surgery including active duty and DoD (Department of Defense) beneficiaries. Prior to being approached for the study, all patients will have had a previous desire for surgery and had a pre-operative evaluation indicating healthy ocular status.

Patients scheduled for PRK surgery will be briefed on the purpose of the study and invited to participate at the preoperative appointment. After the consent process, patients will be randomized in a 1:1 fashion to receive either oral pregabalin 75mg twice daily or placebo for pain control, in addition to the standard care treatment of as needed Percocet and tetracaine ophthalmic drops. Subjects will be evaluated daily for 4 days post-operatively for subjective pain assessment, adverse drug events and compliance, use of concomitant medications as well as monitoring of healing time. Quality of life will be measured at baseline and post-op day 2 when the peak of pain is anticipated. Analysis will be performed to detect an approximate 10% improvement in pain scores. Secondary outcomes will include measuring healing time, quality of life and use of rescue medications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ocular status
* Stable preoperative refractive anisometropia
* Consented to the PRK surgical procedure

Exclusion Criteria:

* Pregnant or breastfeeding
* Diagnosed with autoimmune disease or diabetes
* Patients with a known adverse reaction or hypersensitivity to gabapentin or pregabalin
* Patients only desiring PRK on one eye
* Patients with history of drug use/abuse/addiction
* Patients who are on chronic pain medications
* Patients currently taking anti-epileptic, antidepressant and/or anti-psychotic medications
* Patients with a history of suicidality
* Patients with chronic renal insufficiency (defined as estimated creatinine clearance less than 30ml/min or Scr ≥ 2.0) 10) Patients who have experienced angioedema, or have heart failure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Meek, PharmD, Principal Investigator — 59th Medical Wing; Charles Reilly, MD, Study Chair — 59th Medical Wing; Margaret Bonnie Rosbolt, PharmD, CCRC, Study Director — 59th Medical Wing
Locations (1):
- Wilford Hall Medical Center - Refractive Surgery Center, Lackland Air Force Base, Texas, United States

REFERENCES:
- [Result] Meek JM, Rosbolt MB, Taylor KR, Fusco EA, Panday VA, Reilly CD. Pregabalin versus placebo in postoperative pain relief of patients' status post photorefractive keratectomy: a double-masked, randomized, prospective study. J Ocul Pharmacol Ther. 2014 Sep;30(7):527-32. doi: 10.1089/jop.2013.0208. Epub 2014 Jun 10. PMID 24914779

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: pregabalin: 1 capsule (75 mg) PO BID starting two hours prior to surgery and continuing 4 days postoperatively.
- Lactose Capsule: Placebo: 1 capsule PO BID starting two hours prior to surgery and continuing 4 days postoperatively.
Period: Overall Study
Arm/Group | Pregabalin | Lactose Capsule
Started | 67 | 63
Completed | 67 | 62
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Lactose Capsule | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Mean (Full Range); unit: years] | 34.6 [21 to 57] | 35.1 [21 to 57] | 34.85 [21 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 30 | 30 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 38 | 45 | 83
  Black | 12 | 7 | 19
  Latino | 12 | 11 | 23
  Other | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 67 | 63 | 130

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy
Description: Determine if clinical efficacy is achieved with pregabalin administered prior to PRK and continued for 5 days. This will be evaluated using the short-form McGill pain questionnaire (SF-MPQ). Primary efficacy is assessed on 100mm Visual Analog Scale (VAS); total range is 0 to 100. A score closer to zero indicates a better outcome of less pain.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Lactose Capsule
Number analyzed (Participants) | 67 | 63
units on a scale
  Baseline | 0.89 (2.51) | 1.33 (8.3)
  Surgery Day | 7.56 (10.95) | 10.34 (16.55)
  Postop day 1 morning | 6.32 (9.14) | 10.22 (15.27)
  Postop day 1 evening | 21.32 (21.95) | 27.09 (25.03)
  Postop day 2 morning | 23.49 (21.31) | 29.27 (25.1)
  Postop day 2 evening | 26.14 (22.79) | 25.78 (26.66)
  Postop day 3 morning | 8.48 (12.84) | 8.76 (15.66)
  Postop day 3 evening | 3.48 (6.74) | 6.02 (11.18)
  Postop day 4 morning | 1.9 (4.56) | 2.65 (7.7)
Statistical Analysis 1: Comparison: Pregabalin vs Lactose Capsule; This study was designed to determine if pregabalin is an effective regimen for postoperative pain control following PRK. We hypothesized that there will be at least a 10% improvement in pain after PRK using a scheduled pregabalin dosing regimen compared to placebo. A power analysis was completed to determine the number of patients necessary; Test type: Superiority; p = 0.180, ANOVA

2. Secondary Outcome: PPI Score
Description: Determine if clinical efficacy is achieved with pregabalin administered prior to PRK and continued for 5 days. This will be evaluated using the short-form McGill pain questionnaire (SF-MPQ). Secondary efficacy is assessed with present pain intensity (PPI) score. Scale is 0 (no pain) to 5 (excruciating pain)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Lactose Capsule
Number analyzed (Participants) | 67 | 63
score on a scale
  Baseline | 0.03 (0.17) | 0.03 (0.25)
  Surgery Day | 0.69 (0.76) | 0.84 (0.79)
  Postop day 1 morning | 0.67 (0.73) | 0.89 (0.88)
  Postop day 1 evening | 1.37 (0.89) | 1.62 (1.24)
  Postop day 2 morning | 1.43 (0.89) | 1.62 (0.99)
  Postop day 2 evening | 1.46 (0.94) | 1.48 (1.05)
  Postop day 3 morning | 0.67 (0.77) | 0.68 (0.93)
  Postop day 3 evening | 0.3 (0.58) | 0.48 (0.78)
  Postop day 4 morning | 0.18 (0.46) | 0.22 (0.66)
Statistical Analysis 1: Comparison: Pregabalin vs Lactose Capsule; Test type: Superiority; p = 0.207, ANOVA

3. Secondary Outcome: Total MPQ Score
Description: Determine if clinical efficacy is achieved with pregabalin administered prior to PRK and continued for 5 days. This will be evaluated using the short-form McGill pain questionnaire (SF-MPQ). Secondary efficacy is assessed using the Total MPQ Score. Scale minimum is 0 (no pain) to maximum of 45 (severe pain). A higher score indicates a worse outcome.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Lactose Capsule
Number analyzed (Participants) | 67 | 63
score on a scale
  Baseline | 0.15 (0.47) | 0.16 (0.85)
  Surgery Day | 1.85 (2.28) | 2.18 (3.01)
  Postop day 1 morning | 1.79 (2.16) | 2.16 (2.36)
  Postop day 1 evening | 4.6 (5.07) | 5.37 (6.67)
  Postop day 2 morning | 4.67 (3.9) | 5.61 (6.5)
  Postop day 2 evening | 4.87 (4.1) | 5.68 (7.54)
  Postop day 3 morning | 1.7 (2.34) | 2.9 (6.21)
  Postop day 3 evening | 0.97 (2.02) | 1.16 (1.72)
  Postop day 4 morning | 0.6 (1.35) | 0.39 (1.22)
Statistical Analysis 1: Comparison: Pregabalin vs Lactose Capsule; Test type: Superiority; p = 0.283, ANOVA

4. Secondary Outcome: Quality of Life - BPI
Description: Determine if there was an improvement in the patient's functional health and well-being associated with pregabalin compared to standard of care as assessed by Brief Pain Inventory-short form (BPI-SF). Data was assessed on the day of surgery (Day 0) and at the expected peak of pain, postop Day 2 in the morning. Scale is minimum 0 (no pain) to maximum of 10 (pain as bad as you can imagine). A higher score indicates a worse outcome.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Lactose Capsule
Number analyzed (Participants) | 67 | 63
score on a scale
  Pain at its Worst, Day0 | 0.51 (1.02) | 0.24 (1.011)
  Pain at its Worst, Day2 | 3.76 (2.511) | 4.67 (2.84)
  Pain at its Least, Day 0 | 0.13 (0.519) | 0.08 (0.517)
  Pain at its least, Day2 | 1.31 (1.588) | 1.48 (1.83)
  Avg Pain, Day0 | 0.37 (0.693) | 0.33 (1.122)
  Avg Pain, Day2 | 2.28 (1.929) | 3.03 (2.155)
  Pain Interference, Day0 | 0.13 (0.484) | 0.13 (0.742)
  Pain Interference, Day2 | 2.56 (2.161) | 3.5 (2.832)
Statistical Analysis 1: Comparison: Pregabalin vs Lactose Capsule; Test type: Superiority — Question 1: Pain at its worst; p = 0.223, ANOVA

5. Secondary Outcome: Clinical Efficacy 2
Description: Determine if there was a reduction in the need for use of rescue pain medications, Percocet and tetracaine, in those subjects who received pregabalin. Total number of doses was collected. A higher number of doses required indicates a worse outcome.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Rescue medication doses
Arm/Group | Pregabalin | Lactose Capsule
Number analyzed (Participants) | 67 | 63
Rescue medication doses
  Surgery Day | 0.81 (1.234) | 0.94 (1.134)
  Postop Day 1 | 1.7 (1.842) | 2.44 (2.014)
  Postop Day 3 | 1.7 (1.633) | 2.56 (2.589)
  Postop Day 4 | 0.43 (0.802) | 0.62 (1.25)
Statistical Analysis 1: Comparison: Pregabalin vs Lactose Capsule; Test type: Superiority; p = 0.311, ANOVA

6. Secondary Outcome: Epithelial Healing Time
Description: Determine if there was a reduction in healing time associated with pregabalin as seen with daily slit-lamp observation. Epithelial defect was measured at post-operative day 3, 5, 7, and 9 in each eye. A higher number of days required for healing indicates a worse outcome.
Time Frame: 5 days or more
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: eyes
Arm/Group | Pregabalin | Lactose Capsule
Number analyzed (Participants) | 67 | 63
Number analyzed (eyes) | 134 | 126
Days
  Days to Heal OD (Right Eye) | 3 (1.087) | 2.9 (0.856)
  Days to Heal OS (Left Eye) | 3.09 (1.164) | 2.9 (0.856)
Statistical Analysis 1: Comparison: Pregabalin vs Lactose Capsule; Days to Heal, OD; Test type: Superiority; p = 0.581, t-test, 2 sided
Statistical Analysis 2: Comparison: Pregabalin vs Lactose Capsule; Days to Heal, OS; Test type: Superiority; p = 0.307, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5 days
Description: Adverse events were self-reported by the patients to the investigators at each follow-up evaluation.
  Each adverse event reported was monitored daily until resolution.
Arm/Group | Pregabalin | Lactose Capsule
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/62
Other Adverse Events (participants affected / at risk) | 29/67 | 13/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=67) | Lactose Capsule (N=62)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (11)
Somnolence (Nervous system disorders) | 9 (9) | 0 (0)
Dizziness/Lightheadedness (Nervous system disorders) | 10 (10) | 2 (2)
Rhinorrhea/congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes